CLINICAL TRIAL: NCT06821425
Title: Melatonin Gel as an Adjunct to Xenograft in the Surgical Management of Intrabony Periodontal Defects (A Randomized Controlled Clinical Study)
Brief Title: Melatonin Gel as an Adjuvant in the Surgical Management of Intrabony Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Muhammad Abdelnasser Ali Elnaggar, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-RecIM122330
Record Dates: First submitted 2025-01-08; First posted 2025-02-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Disease, AVDC Stage 3
Keywords: Stage III periodontitis; Melatonin gel; Xenograft
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin gel with Xenograft group (Experimental): Ten patients with stage III periodontitis with vertical bone defects will be subjected to application of particulate xenograft mixed with 5% melatonin gel.
  Interventions: Drug: Melatonin gel mixed with xenograft
- Xenograft Only group (Active Comparator): Ten patients with stage III periodontitis with vertical bone defects will be subjected to application of particulate xenograft alone.
  Interventions: Other: Xenograft

INTERVENTIONS:
Drug: Melatonin gel mixed with xenograft — This study will be conducted to evaluate the effect of melatonin (5% gel) when used as an adjunct to xenograft for the surgical management of intrabony periodontal defects.
  Arms: Melatonin gel with Xenograft group
Other: Xenograft — Application of Xenograft alone for the surgical management of intrabony periodontal defects.
  Arms: Xenograft Only group

SUMMARY:
Surgical periodontal therapy is a commonly employed treatment approach aimed at arresting disease progression and promoting tissue regeneration. Despite advancements in surgical techniques, adjunctive therapies are being explored to enhance the outcomes of periodontal surgical debridement. Melatonin, a hormone primarily known for its role in regulating the sleep-wake cycle, has emerged as a promising candidate for periodontal therapy. It possesses potent antioxidant, anti-inflammatory, and immunomodulatory properties, which make it an attractive therapeutic agent for treating periodontitis. Additionally, melatonin has been linked to bone metabolism, with evidence suggesting its involvement in bone formation and remodeling processes. Bone regeneration is a vital aspect of periodontal therapy, as the restoration of lost osseous structures is crucial for long-term stability of affected teeth. Previous studies have suggested that melatonin may exert positive effects on bone formation by promoting osteoblast differentiation, stimulating matrix synthesis, and inhibiting osteoclast activity. However, limited research has been conducted to specifically evaluate its influence on bone regeneration in the context of surgical periodontal flap therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders within age range of 35-55 years.
2. Patients diagnosed with periodontitis Stage III (Caton et al., 2018; Papapanou et al., 2018).

   Test site criteria: (probing pocket depth ≥6mm and CAL ≥5mm and 3-wall intrabondy defect). All these criteria will be determined after phase I conventional periodontal therapy.
3. Patients with three-wall intrabony defects.
4. Systemically free patients as evidenced by Burket's oral health history questionnaire (Glick et al., 2008)
5. Ability to attend the treatment sessions and comply with the procedures, recall visits and oral hygiene measures.

Exclusion Criteria:

1. Smokers. (Reynolds et al., 2015)
2. Drug abusers.
3. Pregnant or lactating females.
4. Patients under any medication that affect periodontal healing.
5. Vulnerable individuals.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
- Radiographic evaluation of the changes in the intrabony defect | 6 months
  The amount of bone gain in millimeters in follow up radiograph compared to preoperative radiograph

SECONDARY OUTCOMES:
Clinical evaluation of the changes in periodontal parameters | Baseline and 6 months
  The amount of reduction in Probing pocket depth (PD) in mm The new level of clinical attachment (CAL) in relation the CEJ in mm
Evaluation of surgical wound healing | 1 and 2 weeks after surgery.
  Early Healing Index (EHI) to assess the quality of a wound in the days or weeks following a procedure, developed by Wachtel et al. to evaluate flap closure, the presence and amount of fibrin (a blood clot component), and the degree of tissue necrosis. A lower EHI score (such as 1-3) indicates better, complete healing, whereas higher scores (e.g., 4-5) suggest incomplete or poor healing.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided